CLINICAL TRIAL: NCT00626106
Title: An International, Randomized, Double-blind, Placebo-controlled, Phase 2 Study of AMG 479 With Exemestane or Fulvestrant in Postmenopausal Women With Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: QUILT-2.015: A Study of AMG 479 With Exemestane or Fulvestrant in Postmenopausal Women With Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060362; QUILT-2.015 (Other: NantCell, Inc.)
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2016-10

CONDITIONS: Breast Cancer; Breast Tumors; Metastatic Cancer
Keywords: postmenopausal; hormone receptor positive; locally advanced; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — ganitumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy (Active Comparator)
  Interventions: Drug: AMG 479
- Arm B: placebo IV Q2W + Endocrine Therapy (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 479 — AMG 479 administered with exemestane or fulvestrant
  Arms: Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy
Drug: Placebo — Placebo administered with either exemestane or fulvestrant
  Arms: Arm B: placebo IV Q2W + Endocrine Therapy

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase 2 study. Subjects will include postmenopausal women with confirmed HR-positive, locally advanced or metastatic breast cancer, who have disease progression during or within 12 months after completing prior adjuvant endocrine therapy or during the first prior endocrine therapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma of the breast with locally advanced or metastatic disease
* Confirmation of hormone receptor (HR) positive disease status
* Amenable to receive endocrine therapy
* Disease progression while receiving prior endocrine therapy for locally advanced or metastatic breast cancer
* Postmenopausal woman ≥ 18 years old

Exclusion Criteria:

* HR-unknown or HR-negative disease
* Not amenable to endocrine therapy
* Central nervous system metastasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2008-03-27 (Actual); Primary Completion 2010-05-05 (Actual); Study Completion 2011-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (58):
- United States (25):
  - Research Site, Chandler, Arizona
  - Research Site, Anaheim, California
  - Research Site, Beverly Hills, California
  - Research Site, Concord, California
  - Research Site, Duarte, California
  - Research Site, Montebello, California
  - Research Site, San Francisco, California
  - Research Site, Sylmar, California
  - Research Site, Stamford, Connecticut
  - Research Site, Boca Raton, Florida
  - Research Site, Boynton Beach, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Lebanon, New Hampshire
  - Research Site, Denville, New Jersey
  - Research Site, High Point, North Carolina
  - Research Site, Hershey, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, American Fork, Utah
  - Research Site, Tacoma, Washington
- Australia (5):
  - Research Site, Waratah, New South Wales
  - Research Site, Woodville South, South Australia
  - Research Site, Footscray, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Malvern, Victoria
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Ottawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- France (8):
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Reims
  - Research Site, Saint-Herblain
- Germany (3):
  - Research Site, Frankfurt
  - Research Site, Hanover
  - Research Site, Munich
- Research Site, Dublin, Ireland
- Spain (4):
  - Research Site, Barcelona, CataluÃ±a
  - Research Site, L'Hospitalet de Llobregat, CataluÃ±a
  - Research Site, Sabadell, CataluÃ±a
  - Research Site, Madrid
- Switzerland (3):
  - Research Site, Chur
  - Research Site, Lucerne
  - Research Site, Zurich
- United Kingdom (4):
  - Research Site, Derby
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Peterborough

REFERENCES:
- [Background] Robertson JF, Ferrero JM, Bourgeois H, Kennecke H, de Boer RH, Jacot W, McGreivy J, Suzuki S, Zhu M, McCaffery I, Loh E, Gansert JL, Kaufman PA. Ganitumab with either exemestane or fulvestrant for postmenopausal women with advanced, hormone-receptor-positive breast cancer: a randomised, controlled, double-blind, phase 2 trial. Lancet Oncol. 2013 Mar;14(3):228-35. doi: 10.1016/S1470-2045(13)70026-3. Epub 2013 Feb 13. PMID 23414585
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
Started | 106 | 50
Completed | 39 | 26
Not Completed | 67 | 24
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 4
Not completed — Death | 64 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy | Total
Number analyzed (Participants) | 106 | 50 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.4) | 61.7 (10.2) | 62.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 50 | 156
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 106 | 49 | 155
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 100 | 47 | 147
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Postmenopausal Women with Hormone Receptor Positive Locally Advanced or Metastatic Breast Cancer [Count of Participants; unit: Participants] | 106 | 50 | 156

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first observation of disease progression (as classified by modified RECIST), symptomatic deterioration or death due to any cause, whichever occurs first. Disease progression per RECIST is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: Subject completing study will be contacted by the study staff by telephone or at routine clinic visits approximately every 3 months, up to approximately 3 years and 6 months.
Measure: Median (80% Confidence Interval); unit: Months
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
Number analyzed (Participants) | 106 | 50
Months | 3.9 [3.6 to 5.3] | 5.7 [4.4 to 7.4]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Graded Using the National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events(CTCAE) Version 3.0
Time Frame: 30 days after the last dose of study treatment, up to 109 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
Number analyzed (Participants) | 106 | 50
Participants | 105 | 47

3. Secondary Outcome: Cmax of AMG 479
Description: Serum AMG 479 Concentrations After IV Administration of 12 mg/kg AMG 479 in combination with Exemestane, and in combination with Fulvestrant (Cmax).
Time Frame: as for outcome 1
Population: PK population, included only subjects who received the specified combination.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy
Number analyzed (Participants) | 70
μg/mL
  AMG 479 in combination with Exemestane, Cycle 1 Day 1 | 231 (61.8)
  AMG 479 in combination with Exemestane, Cycle 2 Day 1 | 257 (66.9)
  AMG 479 in combination with Exemestane, Cycle 3 Day 1 | 289 (52.7)
  AMG 479 in combination with Fulvestrant, Cycle 1 Day 1 | 225 (46.3)
  AMG 479 in combination with Fulvestrant, Cycle 2 Day 1 | 267 (79.3)
  AMG 479 in combination with Fulvestrant, Cycle 3 Day 1 | 268 (66.7)

4. Secondary Outcome: Clinical Benefit and Objective Response Rate
Description: Clinical benefit was defined as complete/partial response, or stable disease≥24 weeks per modified RECIST/local review.
  Objective response rate was defined as complete/partial response per modified RECIST/local review.
  Per Response Evaluation Criteria in Solid Tumors [RECIST]: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease is disease that is not complete, partial or progressive (PD = at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study)
Time Frame: as for outcome 1
Population: All Randomized Subjects with Baseline Tumor Assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
Number analyzed (Participants) | 63 | 32
Participants
  Objective Response Rate | 5 | 4
  Clinical Benefit Rate | 22 | 10

5. Secondary Outcome: Duration of Response and Time-to-response
Description: Duration of response was defined as time from the date of first confirmed response to the date of first disease progression or death due to any cause in a subset of subjects with confirmed response.
  Time to response was defined as the interval in days from randomization to the first assessment of objective response (CR or PR).
  A complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease is at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study.
Time Frame: as for outcome 1
Population: Subjects with Baseline Measureable Disease and Confirmed Response
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
Number analyzed (Participants) | 5 | 4
Weeks
  Time to Response | 22.1 (13.1) | 19.5 (13.6)
  Duration of Response | 26.5 (10.6) | 31.7 (19.0)

6. Secondary Outcome: Time To Progression, Time-to-treatment Failure, Overall Survival
Description: Time to progression was defined as the time from date of randomization to the date of first occurrence of disease progression or death due to disease progression
  Time to treatment failure was defined as the time from date of randomization to the earliest date of disease progression, death, or end of cycle [last dose date + 1 cycle time: 14 days] for the last dose of ganitumab or placebo regardless of the reason of discontinuation
  Overall survival was defined as the time from randomization to death.
  Progressive disease is at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study.
Time Frame: as for outcome 1
Measure: Median (80% Confidence Interval); unit: Weeks
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
Number analyzed (Participants) | 106 | 50
Weeks
  Time To Progression | 17.0 [15.9 to 23.1] | 24.6 [19.0 to 32.0]
  Time-to-treatment failure | 15.8 [14.0 to 20.0] | 21.6 [18.6 to 31.4]
  Overall Survival | 96.6 [82.3 to NA] — N/A = Not estimable due to insufficient number of participants with events | NA [82.6 to NA] — N/A = Not estimable due to insufficient number of participants with events

7. Secondary Outcome: Global Health Status Time-Adjusted AUC
Description: Based on the European Organization Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ C-30) v3, a 30-item questionnaire comprised of 5 functional scales, 3 symptom scales, and 6 single item scales, all with scores ranging from 1=not at all to 4=very much, along with the Health-Related Quality of Life scale with scores ranging from 1=very poor to 7=excellent; and 2 questions from the Dermatology Life Quality Index (DLQI; scores ranged from 1=not at all to 4=very much). Summing of all these questions and standardizing yielded a total score ranging from 0-100; higher total scores = better quality of life.
  AUC of the change from baseline of the mean total score over time were calculated using the linear trapezoidal rule. The time-adjusted AUC was calculated by dividing the AUC by the time interval between baseline and the last scheduled assessment, the difference was analyzed using analysis of covariance with baseline score and stratification factors as covariates.
Time Frame: From start of study, on Day 1 of cycles 2, 3, and 4 and Day 1 every 3rd cycle thereafter, up to cycle 25 (Cycle = 28 days), approximately 700 days.
Population: The European Organization for Research and Treatment of Cancer (EORTC) analysis set consisted of all subjects in the full analysis set who had a baseline and at least
  1 postbaseline non-missing measurable score of the EORTC QLQ-C30 questionnaire for descriptive comparisons between treatment groups.
Measure: Mean (Full Range); unit: scores*day
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
Number analyzed (Participants) | 95 | 45
scores*day | 1.56 [0.55 to 1.95] | 1.59 [1.18 to 1.95]
Statistical Analysis 1: Comparison: Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy vs Arm B: Placebo IV Q2W + Endocrine Therapy; Test type: Superiority; p = 0.542, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.11 to 0.07]

ADVERSE EVENTS:
Time Frame: 30 days after the last dose of study treatment, up to 109 weeks
Description: Mortality was measured for all subjects, adverse events were measured for the safety population (all subjects who received at least 1 dose of treatment).
Arm/Group | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy | Arm B: Placebo IV Q2W + Endocrine Therapy
All-Cause Mortality (participants affected / at risk) | 64/106 | 19/50
Serious Adverse Events (participants affected / at risk) | 27/106 | 9/49
Other Adverse Events (participants affected / at risk) | 105/106 | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy (N=106) | Arm B: Placebo IV Q2W + Endocrine Therapy (N=49)
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 2 | 1
Asthenia (General disorders) | 2 | 0
Chest Pain (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Campylobacter Intestinal Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Pneumonia (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary Tract Infection Enterococcal (Infections and infestations) | 1 | 0
Migraine (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Horner's Syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: AMG 479 12 mg/kg IV Q2W + Endocrine Therapy (N=106) | Arm B: Placebo IV Q2W + Endocrine Therapy (N=49)
Nausea (Gastrointestinal disorders) | 42 | 19
Diarrhoea (Gastrointestinal disorders) | 33 | 14
Vomiting (Gastrointestinal disorders) | 23 | 10
Constipation (Gastrointestinal disorders) | 16 | 9
Abdominal Pain (Gastrointestinal disorders) | 12 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 5
Stomatitis (Gastrointestinal disorders) | 6 | 1
Fatigue (General disorders) | 42 | 12
Asthenia (General disorders) | 24 | 18
Pyrexia (General disorders) | 12 | 4
Mucosal Inflammation (General disorders) | 12 | 3
Chills (General disorders) | 10 | 3
Oedema Peripheral (General disorders) | 7 | 5
Chest Pain (General disorders) | 6 | 4
Pain (General disorders) | 6 | 2
Infusion Related Reaction (General disorders) | 6 | 1
Injection Site Pain (General disorders) | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 20 | 12
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 17 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 15 | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 12 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 10 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Neck Pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 6 | 0
Headache (Nervous system disorders) | 25 | 13
Dizziness (Nervous system disorders) | 11 | 4
Dysgeusia (Nervous system disorders) | 7 | 3
Paraesthesia (Nervous system disorders) | 5 | 4
Sciatica (Nervous system disorders) | 6 | 3
Tremor (Nervous system disorders) | 5 | 2
Migraine (Nervous system disorders) | 2 | 4
Somnolence (Nervous system disorders) | 1 | 5
Rash (Skin and subcutaneous tissue disorders) | 20 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 8 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8 | 2
Nail Disorder (Skin and subcutaneous tissue disorders) | 6 | 0
Nasopharyngitis (Infections and infestations) | 6 | 6
Urinary Tract Infection (Infections and infestations) | 7 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 2
Sinusitis (Infections and infestations) | 8 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 16 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 0
Hot Flush (Vascular disorders) | 12 | 12
Hypertension (Vascular disorders) | 6 | 5
Insomnia (Psychiatric disorders) | 12 | 8
Anxiety (Psychiatric disorders) | 11 | 6
Depression (Psychiatric disorders) | 7 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 1
Anaemia (Blood and lymphatic system disorders) | 9 | 4
Neutropenia (Blood and lymphatic system disorders) | 11 | 1
Weight Decreased (Investigations) | 9 | 2
Contusion (Injury, poisoning and procedural complications) | 8 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 5
Hypersensitivity (Immune system disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-06-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT00626106/Prot_SAP_000.pdf